CLINICAL TRIAL: NCT01153035
Title: ABLATE Registry: Radiofrequency Ablation After Breast Lumpectomy (eRFA) Added To Extend Intraoperative Margins in the Treatment of Breast Cancer
Brief Title: Excision Followed by Radiofrequency Ablation for Breast Cancer
Acronym: ABLATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104603; NCT01420380 (obsolete NCT alias)
Record Dates: First submitted 2010-06-24; First posted 2010-06-29 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast Conservation Therapy; Lumpectomy; Radiofrequency Ablation; Radiation
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiofrequency Ablation

ARMS (1):
- Surgery followed by RFA (Other)
  Interventions: Device: Radiofrequency Ablation

INTERVENTIONS:
Device: Radiofrequency Ablation — Breast conservation surgery followed by Radiofrequency Ablation of the cavity
  Other Names: AngioDynamics, Inc.

SUMMARY:
The purpose of this study will be to evaluate, in a multi-center setting, the ability of radiofrequency ablation (RFA) of breast cancer lumpectomy sites to extend the "final" negative margin and consequently decrease the rates of re-operation. During the initial breast conservation procedure (lumpectomy), immediately following routine surgical resection of the tumor, radiofrequency energy (RFA) is applied to the wall (bed) of the fresh lumpectomy cavity, thus extending tumor free margin radially beyond the volume of the resected specimen.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a female, ≥ 50 years of age
* The tumor size is ≤ 3 cm (on pre-study radiologic OR clinical exam)
* The tumor is unicentric and unilateral
* The tumor is not involving the skin
* Pathology confirms ductal in situ (DCIS) OR infiltrating ductal carcinoma (IDC), grade I-III
* If tumor is IDC, pathology must be hormone receptor positive (ER+ and/or PR+)
* Patient signs current written informed consent and HIPAA forms

Exclusion Criteria:

* Patient is under 50 years of age
* Patient is male
* Tumor > 3 cm in diameter
* Bilateral malignancy
* Clinically positive lymph nodes
* Tumor involving the skin
* Pathology confirms invasive lobular carcinoma
* Breast implants
* Less than 2 years disease-free survival from previous breast cancer
* Neoadjuvant chemotherapy or chemotherapy for another breast cancer within two years

Ages: 50 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-06; Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Estimate the re-excision rate for close (<3mm) or positive margins | Post-surgery (defined as 2 weeks after surgery, to allow time for pathology to be completed)
  How many patients must go back for re-excision of margins
Decrease local recurrence | Monitor throughout 5 year follow-up
  The patient will be followed closely from the time of surgery through a period of 5 years in order to assess the frequency of local recurrence, defined as a new diagnosis of cancer at or near the site of primary surgery. It is our thought that the addition of RFA to the standard surgical treatment will reduce the number of local recurrences.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ochoa, MD, Principal Investigator — University of Arkansas
Locations (6):
- United States (6):
  - University of Arizona, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sharp Oncology (Comprehensive Breast Care of San Diego), San Diego, California
  - Comprehensive Breast Care of Denver, Denver, Colorado
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Columbia, New York, New York

REFERENCES:
- [Background] Klimberg VS, Ochoa D, Henry-Tillman R, Hardee M, Boneti C, Adkins LL, McCarthy M, Tummel E, Lee J, Malak S, Makhoul I, Korourian S. Long-term results of phase II ablation after breast lumpectomy added to extend intraoperative margins (ABLATE l) trial. J Am Coll Surg. 2014 Apr;218(4):741-9. doi: 10.1016/j.jamcollsurg.2013.12.032. Epub 2014 Jan 11. PMID 24655863
- [Result] Mackey A, Feldman S, Vaz A, Durrant L, Seaton C, Klimberg VS. Radiofrequency ablation after breast lumpectomy added to extend intraoperative margins in the treatment of breast cancer (ABLATE): a single-institution experience. Ann Surg Oncol. 2012 Aug;19(8):2618-9. doi: 10.1245/s10434-012-2293-7. Epub 2012 Mar 16. PMID 22422482
- [Result] Wilson M, Korourian S, Boneti C, Adkins L, Badgwell B, Lee J, Suzanne Klimberg V. Long-term results of excision followed by radiofrequency ablation as the sole means of local therapy for breast cancer. Ann Surg Oncol. 2012 Oct;19(10):3192-8. doi: 10.1245/s10434-012-2476-2. Epub 2012 Aug 22. PMID 22911363